CLINICAL TRIAL: NCT00216593
Title: Treatment of Severe Alzheimer's Disease in a Residential Home, Nursing Home, or Geriatric Residential Setting: Evaluation of Efficacy and Safety of Galantamine Hydrobromide in a Randomised, Doubleblind, Placebo-Controlled Study.
Brief Title: Treatment of Severe Alzheimer's Disease: Evaluation of Efficacy and Safety of Galantamine Hydrobromide in a Controlled Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003940
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2010-04

CONDITIONS: Dementia; Alzheimer Disease
Keywords: dementia; cognition function; Alzheimer disease; behavioral symptoms; galantamine hydrobromide
MeSH Terms: conditions — Dementia; Alzheimer Disease; Behavioral Symptoms | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of galantamine hydrobromide treatment in patients with severe Alzheimer's disease.

DETAILED DESCRIPTION:
This is a multicenter, 1-year study that includes a randomized, 6-month, double-blind, placebo-controlled phase and a 6-month open-label extension of galantamine hydrobromide treatment in subjects with severe Alzheimer's disease. The open-label extension is optional for al patients. Patients eligible for the study will be randomized to treatment with either galantamine hydrobromide or placebo over 6 months for the first phase of the study. The principal measures include the results of the Severe Impairment Battery and the Minimum Data Set-Activities of Daily Living tests, to assess aspects of cognition and behavior, and impact on the patient's ability to perform normal daily activities. Additional evaluations include the Neuro-Psychiatric Inventory-Nursing Home Version measure and 2 subscales of the Minimum Data Set tests to further assess patients behavior, social and physical functioning, the level of caregiver support needed, and impact to the patient's caregiver; the Mini-Mental State Examination, to assess cognitive abilities; and external health-and social-service use. Safety and tolerability will be evaluated on the basis of adverse event reports, physical examination, electrocardiograms, vital signs, and laboratory parameters. The study hypothesis is that treatment with galantamine, compared with placebo, will significantly improve cognition and ability to function in patients with severe Alzheimer's disease, and is generally well-tolerated. Galantamine hydrobromide tablets taken by mouth two times daily: 4 weeks at 8 milligrams (mg)/day, 4 weeks at 16 mg/day, increased to 24 mg/day for the remainder of the 6 months. Dose may be reduced at investigator's discretion. Galatamine hydrobromide for additional 6 months in open-label phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's type dementia, rated as severe
* progressive worsening of memory and other cognitive functions
* brain imaging (CTor MRI scan) within last 3 years
* ability to be mobile (aided or unaided) with sufficient vision and hearing to comply with testing.

Exclusion Criteria:

* Dementia caused by cerebrovascular disease
* disturbances of consciousness, delirium, psychosis
* severe aphasia
* or major sensorimotor impairment
* cognitive impairment due to acute cerebral trauma, hypoxic cerebral damage, vitamin deficiency, infections, primary of metastatic cerebral neoplasia, endocrine or metabolic disease or mental retardation, pregnant or nursing women or those without adequate contraception.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2003-12; Primary Completion 2007-09 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in scores from baseline to week 26 on measuring cognition Severe Impairment Battery test and the Minimum Data Set Activities of Daily Living test.

SECONDARY OUTCOMES:
Results from Neuro Psychiatric Inventory-nursing home version test. Safety assessments include reports of adverse events, physical exam, vital signs, electrocardiograms, and laboratory test results.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- [Derived] Burns A, Bernabei R, Bullock R, Cruz Jentoft AJ, Frolich L, Hock C, Raivio M, Triau E, Vandewoude M, Wimo A, Came E, Van Baelen B, Hammond GL, van Oene JC, Schwalen S. Safety and efficacy of galantamine (Reminyl) in severe Alzheimer's disease (the SERAD study): a randomised, placebo-controlled, double-blind trial. Lancet Neurol. 2009 Jan;8(1):39-47. doi: 10.1016/S1474-4422(08)70261-8. Epub 2008 Nov 29. PMID 19042161